CLINICAL TRIAL: NCT01982552
Title: An Observational Study to Assess Patient Satisfaction and Control of Psoriasis With Calcipotriene/Betamethasone Dipropionate (Taclonex®) Topical Suspension, and Effect on Quality of Life
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: APPEAL
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis Vulgaris
Keywords: Plaque psoriasis; calcipotriene; betamethasone dipropionate; topical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to document quality of life, patient satisfaction, effect on itching, and control of psoriasis vulgaris associated with use of calcipotriene/betamethasone dipropionate (Taclonex®) topical suspension 0.005% / 0.064% for treatment of plaque psoriasis under real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained prior to any study related activities
2. Aged 18 years or above
3. Either sex
4. Any race or ethnicity
5. Attending a hospital outpatient clinic or the private practice of a board-certified dermatologist, dermatology-certified nurse practitioner or physician assistant trained in dermatology
6. Clinical diagnosis of psoriasis vulgaris involving scalp and/or body amenable to treatment with a maximum of 100 g of topical medication per week.
7. Patients who receive a prescription of calcipotriene/betamethasone dipropionate (Taclonex®) topical suspension 0.005% / 0.064% as per an investigator's clinical judgment and in accordance with the US label, and who have access to the medication
8. Able to communicate with the investigator, read and understand English, and understand and comply with the requirements of the study

Exclusion Criteria:

1. Prior treatment with calcipotriene/betamethasone dipropionate (Taclonex®) topical suspension, 0.005%/0.064%.
2. Contraindications or any warnings/precautions according to the US label.
3. Current participation in any other interventional clinical study.
4. Females who are pregnant, breast-feeding, or females of child-bearing potential wishing to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending a hospital outpatient clinic or the private practice of a board-certified dermatologist, dermatology-certified nurse practitioner or physician assistant trained in dermatology
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | 8 weeks
  Mean change from baseline

SECONDARY OUTCOMES:
Visual Analogue Scale for itching | 2 and 8 weeks
  Mean percent change from baseline
Patient Global Assessment (PGA) | 2 and 8 weeks
  Percent of subjects with controlled disease
Dermatology Life Quality Index (DLQI) | 2 weeks
  Mean change from baseline
Treatment Satisfaction Questionnaire for Medication (TSQM)-9 | 2 and 8 weeks
Dermatology Life Quality Index (DLQI) | 2 and 8 weeks
  Percent of patients that have a 5 point or greater change in total score

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, MD, Principal Investigator — Psoriasis Treatment Center of Central New Jersey, East Windsor, NJ
Locations (12):
- United States (12):
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - Center for Dermatology Clinical Research, Fremont, California
  - Academic Alliance Dermatology, Clearwater, Florida
  - Dermatology Associates and Research, Coral Gables, Florida
  - Melissa Knuckles Dermatology, Corbin, Kentucky
  - Grekin Skin Institute, Warren, Michigan
  - Bettencourt Skin Center, Henderson, Nevada
  - Las Vegas Skin and Cancer Clinic, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - Skin Specialty Dermatology, New York, New York
  - Center for Clinical Studies, Webster, Texas
  - West End Dermatology, Richmond, Virginia

REFERENCES:
- See also: Result publication — https://www.ncbi.nlm.nih.gov/pubmed/?term=25607705